CLINICAL TRIAL: NCT06650007
Title: A Multicenter, Randomized, Double-blind, Placebo- Parallel Controlled, Phase III Study to Evaluate the Efficacy and Safety of HRS9531 Injection in Subjects With Type 2 Diabetes， Inadequately Controlled With Diet and Exercise Alone
Brief Title: the Efficacy and Safety of HRS9531 Injection in Subjects With Type 2 Diabetes， Inadequately Controlled With Diet and Exercise Alone
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRS9531-302
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental)
  Interventions: Drug: HRS9531 Injection
- Group B (Placebo Comparator)
  Interventions: Drug: HRS9531 Placebo Injection
- Group C (Experimental)
  Interventions: Drug: HRS9531 Injection
- Group D (Placebo Comparator)
  Interventions: Drug: HRS9531 Placebo Injection

INTERVENTIONS:
Drug: HRS9531 Injection — HRS9531 Injection
  Arms: Group A; Group C
Drug: HRS9531 Placebo Injection — HRS9531 Placebo Injection
  Arms: Group B; Group D

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of HRS9531 compared to placebo in controlling blood glucose levels after 24 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, Age ≥18 years at the time of signing informed consent.
2. Diagnosed with type 2 diabetes mellitus (T2DM) for at least 90 days prior to day of screening.
3. Treatment with Diet and Exercise alone at least 90 days prior to day of screening.
4. 7.5% ≤ HbA1c ≤10.0% at screening.

Exclusion Criteria:

1. Uncontrollable hypertension(with or without antihypertensive treatment) : systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg at screening.
2. Diagnosed or suspected with type 1 diabetes mellitus, special types of diabetes or secondary diabetes.
3. History of significant hematological disorders (e.g., sickle cell disease, hemolytic anemia, myelodysplastic syndrome, etc.) or other conditions causing hemolysis or instability of red blood cells (e.g., malaria, hypersplenism, etc.).
4. Presence of an endocrine disorder or history that may significantly affect bady weight(e.g., Cushing's syndrome, hypothyroidism or hyperthyroidism, except hypothyroidism if thyroid hormone replacement dose has been stable for at least 6 months) ；
5. Severe infection, severe trauma, or moderate-to-major surgery within 1 month before screening.
6. Participated in clinical trials of any drug or medical device within 3 months prior to screening, and participation in clinical trials is defined as signing informed consent and using investigational drugs (including placebo) or investigational medical devices; Or is still in the trial drug within 5 half-lives (whichever is Longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | from baseline to 36 weeks treatment

SECONDARY OUTCOMES:
Proportion of subjects with HbA1c<7.0% and ≤6.5% | from baseline to 36 weeks treatment
Change in FPG | from baseline to 36 weeks treatment
Change in body weight | from baseline to 36 weeks treatment
Proportion of subjects with HbA1c<7.0% and weight loss ≥5% | from baseline to 36 weeks treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided